CLINICAL TRIAL: NCT04107285
Title: A Study of Longitudinal Neurocognitive and Neuroimaging Evaluations for Adult Patients With Lymphoma Receiving CD19 CAR T Cell Therapy
Brief Title: Looking at Cognitive and Brain Changes in People With Lymphoma Receiving CAR-T Therapy
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-268
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma Receiving CAR-T Therapy
Keywords: Neurocognitive Evaluations; Neuroimaging Evaluations; 19-268
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurocognitive evaluation prior to and following CART
  Interventions: Behavioral: neurocognitive evaluations; Diagnostic Test: brain MRIs; Other: Blood samples

INTERVENTIONS:
Behavioral: neurocognitive evaluations — The test battery consists of validated and reliable measures of attention, executive functions and memory.
Diagnostic Test: brain MRIs — Patients will undergo baseline and follow-up research MRIs in the same scanner at MSKCC (3 Tesla scanner (GE, Discovery 750W, USA) with a GEM HNU 24-channel head coil) (total scan duration=15 minutes).
Other: Blood samples — Research blood samples will be collected pre-CAR T infusion; day of CART infusion (day 0), and post-infusion days 7, 14, 21, 28 (+/- 7 days), at start of neurotoxicity, and at 3-4 months and 6-7 months post-CART.

SUMMARY:
The purpose of this study is to learn about possible changes in cognitive (mental) abilities, such as memory skills and concentration, and in brain anatomy (structure) and function, in people with lymphoma receiving CAR-T therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Planned treatment with commercial CD19-specific CAR T cells (axicabtagene ciloleucel, tisagenlecleucel, lisocabtagene maraleucel, or brexacabtagene autoleucel) for lymphoma.
* Patients must have adequate end organ function for CAR T cell therapy

  * Eastern Cooperative Group (ECOG) performance status of 0 to 2
  * Meet cardiac, pulmonary, hematologic, hepatic, and renal requirements for CART therapy as described in corresponding product package insert
* No evidence of central nervous system disease at study entry
* Fluent and able to communicate well enough in English to complete the study assessments and provide informed consent, in the judgment of the consenting professional. o Patients who report that English is not their primary language will be asked the US Census English proficiency question: "How well do you speak English," and the answer "very well" will be required

Exclusion Criteria:

* Signs and/or symptoms of central nervous system cancer (e.g., metastases, leptomeningeal disease) as determined by their physician, medical records, or by a brain MRI, either at the time of enrollment or during the study period.
* Current diagnosis of major Axis I psychiatric disorder (DSM-IV), major depression, bipolar disorder, or schizophrenia, as per medical records or patient report
* History of neurodegenerative disease, or traumatic brain injury with loss of consciousness (>60 minutes), as per medical records or patient report
* A history of epilepsy as per medical records or patient report
* Current ongoing substance abuse and/or history of substance abuse, as per medical records or patient report
* Evidence of visual or auditory impairment that would preclude completion of the assessments, as per medical records or patient report
* Contraindications to MRI examinations as per standard screening guidelines used in the Department of Radiology (i.e., ferromagnetic material or implants, pacemakers or defibrillators, stents, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
changes in neurocognitive functions | 1 year
  correlations of neurocognitive scores with the FACIT-FS (fatigue) scale score The Functional Assessment of Chronic Illness Therapy-Fatigue Subscale, Version 4 (FACITFS V-4 56, is a 13-item questionnaire designed to assess symptoms and concerns specific to the QOL of patients with fatigue [66]. The questionnaire asks respondents to indicate the extent to which each item applied to them over "the past 7 days" using a 5-point Likert-type response format ranging from "0 - Not at all" to "4 - Very much". The 13 items produce the Fatigue Subscale (FS) score (range 0 - 52).
changes in functional connectivity | 1 year
  MRIs

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Santomasso, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm